CLINICAL TRIAL: NCT07369011
Title: A Master Protocol for Phase 3 Randomized, Double-Blind, Placebo-Controlled Studies to Investigate the Efficacy and Safety of Once Weekly Eloralintide in Adult Participants With Moderate to Severe Obstructive Sleep Apnea, and Obesity or Overweight
Brief Title: A Study of Eloralintide (LY3841136) in Participants With Obstructive Sleep Apnea and Obesity or Overweight
Acronym: ENLIGHTEN-3
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 27764; J3R-MC-YDAO (Other: Eli Lilly and Company); J3R-MC-YSA1 (Other: Eli Lilly and Company); J3R-MC-YSA2 (Other: Eli Lilly and Company); 2025-523769-11-00 (EU CTIS Number)
Record Dates: First submitted 2026-01-23; First posted 2026-01-27 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Sleep Apnea, Obstructive; Obesity; Overweight
MeSH Terms: conditions — Sleep Apnea, Obstructive; Obesity; Overweight

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Eloralintide (YSA1) (Experimental): Participants will receive eloralintide subcutaneously (SC)
  Interventions: Drug: Eloralintide
- Placebo (YSA1) (Placebo Comparator): Participants will receive placebo SC
  Interventions: Drug: Placebo
- Eloralintide (YSA2) (Experimental): Participants will receive eloralintide SC
  Interventions: Drug: Eloralintide
- Placebo (YSA2) (Placebo Comparator): Participants will receive placebo SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Eloralintide — Administered SC
  Other Names: LY3841136
  Arms: Eloralintide (YSA1); Eloralintide (YSA2)
Drug: Placebo — Administered SC
  Arms: Placebo (YSA1); Placebo (YSA2)

SUMMARY:
The purpose of the studies is to evaluate the efficacy and safety of eloralintide in participants with moderate-to-severe obstructive sleep apnea and obesity or overweight. YDAO is a master protocol designed to support two independent studies: YSA1 and YSA2. Study YSA1 will include participants who are unable or unwilling to use Positive Airway Pressure (PAP) therapy and study YSA2 will include participants who are on PAP therapy for at least 3 months at time of screening and plan to continue PAP therapy during the study.

Participants will be assigned to the Intervention-Specific Appendix (ISA) that reflects their current PAP usage. Participation in the study will last about 76 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed history of moderate-to-severe OSA
* Have an AHI ≥ 15 on polysomnography (PSG) as part of the study at screening
* Have a BMI ≥27 kg/m2 at screening
* Have a stable body weight (<5% body weight change) for 90 days prior to screening
* Have a history of at least one self-reported unsuccessful dietary effort to reduce body weight

For YSA1 Participants:

* Are unable or unwilling to use PAP therapy

For YSA2 Participants:

* Have been on PAP therapy for at least three consecutive months prior to screening and plan to continue PAP therapy during the study

Exclusion Criteria:

* Have a prior or planned surgical treatment for obesity (liposuction, cryolipolysis, or abdominoplasty allowed if performed >1 year before screening)
* Have a prior or planned endoscopic procedure and/or device-based therapy for obesity (prior device-based therapy acceptable if device removal was more than 6 months prior to screening)
* Any previous or planned surgery for sleep apnea or major ear, nose or throat surgery that still may affect breathing at time of screening
* Have type 1 diabetes, type 2 diabetes, or any other type of diabetes
* Have had within 90 days prior to screening:

  * acute myocardial infarction
  * cerebrovascular accident (stroke)
  * coronary artery revascularization
  * unstable angina, or
  * hospitalization due to congestive heart failure
* Have a history or diagnosis of New York Heart Association Functional Classification Class IV congestive heart failure
* Have taken medications or alternative remedies intended for weight loss within 90 days of screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2028-03 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Percent Change from Baseline in Body Weight | Baseline, Week 64
Change from Baseline in Apnea-Hypopnea Index (AHI) | Baseline, Week 64

SECONDARY OUTCOMES:
Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 64
Percent Change from Baseline in Triglycerides | Baseline, Week 64
Percent Change from Baseline in High Sensitivity C-Reactive Protein (hsCRP) | Baseline, Week 64
Change from Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form Sleep-Related Impairment 8a T-Score | Baseline, Week 64
Achievement of AHI <5 or AHI 5-14 with Epworth Sleepiness Scale (ESS) ≤ 10 | Baseline, Week 64
Percent Change from Baseline in Sleep Apnea Specific Hypoxic Burden (SASHB) | Baseline, Week 64
Number of Participants who Achieve ≥50% decrease in AHI | Baseline, Week 64
Change from Baseline in Body Mass Index (BMI) | Baseline, Week 64
Change from Baseline in Fasting Glucose | Baseline, Week 64
Change from Baseline in ESS Score | Baseline, Week 64
Change from Baseline in Short Form-36 (SF-36 v2) Scores | Baseline, Week 64
Change from Baseline in EQ-5D-5L Scores | Baseline, Week 64
Percent Change from Baseline in Fasting Insulin | Baseline, Week 64
Change from Baseline in Waist Circumference | Baseline, Week 64
Change in Medication Use | Baseline, Week 64
Achievement of Improved Categorical Shift in Patient Global Impression of Severity-Obstructive Sleep Apnea (PGIS-OSA) | Baseline, Week 64
Pharmacokinetics (PK): Maximum Concentration at Steady State (Cmax,ss) | Baseline through Week 64
PK: Area Under the Concentration Versus Time Curve for One Dosing Interval at Steady State (AUC(0-ᴛ)ss) | Baseline through Week 64

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 8 AM - 8 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (122):
- United States (24):
  - Cullman Clinical Trials, Cullman, Alabama
  - Ark Clinical Research, Long Beach, California
  - Collaborative Neuroscience Research, LLC, Los Alamitos, California
  - Artemis Institute for Clinical Research, Riverside, California
  - Care Access - Aurora, Aurora, Colorado
  - Flourish Research - Miami, LLC, Miami, Florida
  - PharmaDev Clinical Research Institute, LLC, Miami, Florida
  - Emerald Coast Neurology - Airport Boulevard, Pensacola, Florida
  - Teak Research Consults, Lawrenceville, Georgia
  - EBGS Clinical Research Center, Snellville, Georgia
  - Care Access - Shreveport 2, Shreveport, Louisiana
  - Flourish Research - Bowie, Bowie, Maryland
  - Revive Research Institute, Inc., Southfield, Michigan
  - Headlands Research-Twin Cities, Maplewood, Minnesota
  - Clayton Sleep Institute - St. Louis - Tesson Ferry Road, St Louis, Missouri
  - Palm Research Center Tenaya, Las Vegas, Nevada
  - The Sleep Spot - Maimonides, Albuquerque, New Mexico
  - Rochester Clinical Research - Buffalo, Buffalo, New York
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Heritage Valley Multispecialty Group, Inc, Beaver, Pennsylvania
  - Bogan Sleep Consultants, Columbia, South Carolina
  - FutureSearch Trials of Neurology, Austin, Texas
  - Sleep Therapy Research Center, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
- Argentina (12):
  - Stat Research S.A., Buenos Aires
  - Centro de Investigaciones Metabólicas (CINME), Buenos Aires
  - Centro Médico Viamonte, Buenos Aires
  - Consultorio de Investigación Clínica EMO SRL, Buenos Aires
  - Centro Medico Dra. Laura Maffei- Investigacion Clinica Aplicada, Buenos Aires
  - Fundación Respirar, Buenos Aires
  - Centro de Investigaciones Clínicas Baigorria, Granadero Baigorria
  - Instituto Médico Río Cuarto, Río Cuarto
  - INECO Neurociencias Oroño, Rosario
  - Instituto Médico Fundación Grupo Colaborativo Rosario Investigación y Prevención Medica, Rosario
  - CIMER Centro Integral de Medicina Respiratoria, San Miguel de Tucumán
  - Centro de Salud e Investigaciones Médicas, Santa Rosa
- Australia (9):
  - Nightingale Research, Adelaide
  - Flinders University, Bedford Park
  - Box Hill Hospital, Box Hill
  - Core Research Group, Brisbane
  - Austin Health - Repatriation Hospital, Heidelberg West
  - Woolcock Institute of Medical Research, Macquarie Park
  - CDH Research Institute Pty Ltd, Maroochydore
  - Gold Coast University Hospital, Southport
  - TrialsWest - Spearwood, Spearwood
- Brazil (10):
  - Instituto de Pesquisa clinica de Campinas, Campinas
  - Centro de Pesquisa Clínica de Marília - CPCLIM, Marília
  - Núcleo de Pesquisa Clínica do Rio Grande do Sul, Porto Alegre
  - CEMER - Centro Médico do Recife, Recife
  - Ruschel Medicina e Pesquisa Clínica, Rio de Janeiro
  - Prognosis Pesquisa Clínica, Santo André
  - CPHosp Medicina, Ensino e Pesquisa (CPQuali), São Paulo
  - BR Trials - Ensaios Clinicos e Consultoria, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
  - Incor - Instituto do Coracao, São Paulo
- Canada (6):
  - MyCliniResearch, Inc., Calgary
  - Alpha Recherche Clinique - Lévis, Lévis
  - Alpha Recherche Clinique, Québec
  - C.I.C. Joliette, Saint-Charles-Borromée
  - Maple Leaf Research, Toronto
  - C.I.C. Mauricie inc., Trois-Rivières
- China (15):
  - China-Japan Friendship Hospital, Beijing
  - The First Hospital of Jilin University, Changchun
  - Sichuan Provincial People's Hospital, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Gansu Provincial Hospital, Lanzhou
  - The First Affiliated Hospital of Henan University of Science &Technology, Luoyang Shi
  - Jiangxi Provincial People's Hospital, Nanchang
  - The Second Affiliated Hospital of Nanchang University, Nanchang
  - The Second Affiliated Hospital of Guangxi Medical University, Nanning
  - Shanghai Sixth People's Hospital, Shanghai
  - ShenZhen People's Hospital, Shenzhen
  - The Third Hospital of Hebei Medical University, Shijiazhuang
  - The Second Affiliated Hospital of Soochow University, Suzhou
  - Wuxi People's Hospital, Wuxi
- Germany (8):
  - CIMS Studienzentrum Bamberg, Bamberg
  - Advanced Sleep Research, Berlin
  - InnoDiab Forschung Gmbh, Essen
  - Siteworks GmbH - Hannover, Hanover
  - Siteworks - Karlsruhe, Karlsruhe
  - Universitätsklinikum Marburg, Marburg
  - RED-Institut GmbH, Oldenburg
  - Somni bene, Schwerin
- India (12):
  - SDS Tuberculosis Research Center & Rajiv Gandhi Institute of Chest Diseases, Bengaluru
  - St. Johns Medical College Hospital, Bengaluru
  - Utkal Institute of Medical Sciences and Hospital, Bhubaneswar
  - Endolife Speciality Hospitals, Guntur
  - KRIMS Hospital, Nagpur
  - All India Institute of Medical Sciences, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - Deenanath Mangeshkar Hospital & Research Centre, Pune
  - All India Institute of Medical Sciences, Raipur
  - All India Institute of Medical Sciences - Rishikesh, Rishikesh
  - Bhakti Vedanta Hospital and Research Institute, Thane
  - Rhythm Heart Institute - A Unit of SLPL, Vadodara
- Japan (10):
  - Juntendo University Hospital, Bunkyō City
  - Fukuoka University Hospital, Fukuoka
  - Social Medical Corporation Sokujinkai Sleep and Mental Health Clinic - Kitahiroshima, Kitahiroshima
  - Kirigaokatsuda Hospital, Kitakyushu
  - Toranomon Hospital, Minatoku
  - Osaka Kaisei Hospital, Osaka
  - KKR Sapporo Medical Center, Sapporo
  - Yoyogi Sleep Disorder Center, Shibuya-ku
  - Nakamura Clinic, Urasoe
  - RESM Respiratory and Sleep Medical Care Clinic, Yokohama
- South Korea (4):
  - Korea University Ansan Hospital, Ansan-si
  - Seoul National University Bundang Hospital, Seongnam
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
- Spain (9):
  - Hospital Universitario de Guadalajara, Guadalajara
  - Hospital Universitari de Santa Maria, Lleida
  - Hospital San Pedro, Logroño
  - Hospital Universitario Ramón y Cajal, Madrid
  - Instituto de Investigaciones del Sueño, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Quiron Infanta Luisa, Seville
  - Hospital Universitario Virgen Del Rocio, Seville
- Taiwan (3):
  - China Medical University Hospital, Taichung
  - National Cheng-Kung Uni. Hosp., Tainan
  - Chang Gung Medical Foundation-Linkou Branch, Taoyuan District

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication or approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal should be approved by an independent review panel and researchers should sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- See also: A Study of Eloralintide (LY3841136) in Participants With Obstructive Sleep Apnea and Obesity or Overweight (ENLIGHTEN-3) — https://trials.lilly.com/en-US/trial/687736